CLINICAL TRIAL: NCT04734080
Title: Effects of Perioperative Dronabinol Use in Total Knee Arthroplasty
Brief Title: Dronabinol in Total Knee Arthroplasty (TKA)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019-1416
Record Dates: First submitted 2021-01-19; First posted 2021-02-02 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Total Knee Arthroplasty; Opioid Use
Keywords: Knee Arthroplasty; Dronabinol; Opioid
MeSH Terms: interventions — Dronabinol; Capsules

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Throughout cannabinoid research, there has been concern about potential unblinding due to the side effect profile of this class of medication. Prior meta-analyses have advocated for the use of active placebo, with concern that unblinding may misrepresent the effects of clinical trials. However, due to evidence of histamine receptor involvement in pain transmission, as well as overlap in antihistamine antiemetic use and common cannabinoid side effect profiles, we have chosen to use non-active placebo. Our hope is to elicit maximum benefit of cannabinoid dosing perioperatively without confounding variables. With use of non-active placebo, we will perform a comprehensive blinding analysis following the study period to ensure adequate blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dronabinol (Experimental): 57 subjects undergoing primary Total Knee Arthroplasty will be randomized to receive BID (2x/day) dosing of 5 mg of Dronabinol beginning on the day of surgery and with the final dose on the morning of POD (postoperative day) 2.
  Interventions: Drug: Dronabinol 5mg Cap
- Placebo (Placebo Comparator): 57 subjects undergoing primary Total Knee Arthroplasty will be randomized to receive BID (2x/day) dosing of a non-active placebo pill beginning on the day of surgery and with the final dose on the morning of POD (postoperative day) 2.
  Interventions: Other: Placebo oral tablet

INTERVENTIONS:
Drug: Dronabinol 5mg Cap — Dronabinol is a synthetic tetrahydrocannabinol (THC) agent approved for nausea and vomiting with chemotherapy and as an appetite stimulant in AIDS patients.
  Other Names: marinol
  Arms: Dronabinol
Other: Placebo oral tablet — Non-active placebo
  Other Names: placebo
  Arms: Placebo

SUMMARY:
The goal of this double-blinded randomized controlled trial is to compare whether the addition of Dronabinol compared to a placebo will affect opioid intake in patients undergoing a total knee arthroplasty. The main question it aims to answer are:

1. Does perioperative dronabinol use (starting in the immediate preoperative period (enrollment before 1 PM), with BID dosing concluding the evening of POD2) affect postoperative opioid consumption 24-48 hours following total knee arthroplasty?
2. Is there an effect of perioperative dronabinol use in the total knee arthroplasty patient on POD2 pain scores with ambulation?
3. Will hospital length of stay following total knee arthroplasty be affected in patients who use perioperative dronabinol as compared to control?
4. Does the use of perioperative dronabinol affect time to reach physical therapy discharge goals in postoperative total knee arthroplasty patients?
5. Is there a change in number of postoperative oxygen desaturation events in patients following total knee arthroplasty based on perioperative dronabinol use?

Participants will:

* Be randomized to take the dronabinol or placebo medication in 5 dosage
* Answer survey questions in regard to pain, postop nausea/vomiting, cognitive/adverse event, and outcome quality and support of decision making.
* Be connected to a Masimo to record oxygen saturation and an Actigraph to record sleep quality.

Researchers will compare two groups: 1) intervention group and 2) control group to see if dronabinol affect postoperative opioid consumption 24-48 hours following their total knee arthroplasty surgery.

DETAILED DESCRIPTION:
The objective of this study is to examine the possible therapeutic advantages of administering perioperative dronabinol to individuals who are undergoing unilateral total knee arthroplasty (TKA). With the utilization of contemporary regional anesthetic procedures and peripheral nerve blocks, pain management is typically effective in the immediate aftermath of total knee arthroplasty (TKA) within the first day after surgery. Rebound pain is shown to occur on the second day following postoperative discharge (POD2), once the analgesic blocks administered during the procedure have ceased to be effective. Previous studies have suggested that dronabinol, a synthetic form of THC, may have potential analgesic properties. Our goal is to find out if giving dronabinol before surgery could lower the number of opioids that people need on postoperative day 2 (POD2) in people who are having total knee arthroplasty (TKA). This research could provide valuable insights into alternative pain management strategies for TKA patients, potentially minimizing opioid-related side effects and improving overall patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18-70 years old with osteoarthrosis scheduled for primary unilateral knee arthroplasty with a participating surgeon
* Planned use of regional anesthetic technique during surgery involving infiltration between the popliteal artery and the capsule of the posterior knee (IPACK), adductor canal block (ACB) and periarticular injection (PAI)
* Ability to follow study protocol

Exclusion Criteria:

* Patients less than 18 years of age or older than 70 years of age
* Contraindication to regional or neuraxial anesthetic
* Intended use of general anesthesia
* Revision surgery
* Chronic opioid use (for >3 months prior to surgery)
* Cannabis/cannabinoid use within the last 3 months
* ASA class of IV or greater
* Active or history of major mental history (as defined by the Diagnostic and Statistical Manual of Mental Disorders-5 [DSM-5]; i.e. major depressive disorder, anxiety, bipolar disorder, schizophrenia)
* History of seizures
* Use of antidepressants
* Use of anticonvulsants
* Use of Coumadin
* Use of Disulfuram
* Use of Metronidazole
* Non-English speakers
* BMI ≥40

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Cumulative Opioid Consumption 24-48 hours post-operatively | 24-48 hours post-operatively
  The primary outcome of the study will be cumulative patient opioid consumption 24-48 hours post operatively, defined by total morphine equivalents (MEs). This outcome will be measured throughout the patient hospitalization and conclude at 48 hours after anesthesia stop time.

SECONDARY OUTCOMES:
Time to reach discharge from physical therapy | Post operative day 0 (beginning in the PACU)-Discharge, assessed up to 7 days
  Time to reach discharge physical therapy goals, as defined by the number of hours required to meet the following criteria: stable vital signs during Physical therapy (PT), safe independent transfer from bed to standing as well as transfer in and out of seated position, ability to walk 40 feet only with aid of crutch or walker. This outcome will be measured prior to patient discharge.
Average pain score with ambulation reported on a numeric rating scale (NRS) | Post operative day 1, 3, 7, 90 and 180
  Patient pain with ambulation on POD1, 2, 7, 90 and 180, defined by patient reported Numeric Rating Scale (NRS) pain score, (from 0-no pain to 10-worst pain imaginable).
Average pain score at rest reported on a numeric rating scale (NRS) | Post operative day 0 (beginning in the PACU), POD 1, 2, 7, 90 and 180
  Patient pain at rest upon PACU entry and in the morning of POD1, POD2, POD7, POD90 and POD180 defined by patient reported Numeric Rating Scale (NRS) pain score, (from 0-no pain to 10-worst pain imaginable).
Length of hospital stay (hours) | Post operative day 0 (beginning in the PACU)-Discharge, assessed up to 7 days
  Hospital length of stay from procedure start time to time of discharge
Percentage of time and total time of desaturation events | Post operative day 0 (beginning in the PACU)-48 hours post operative discharge
  Postoperative oxygen desaturation events will be reported in minutes. This outcome will be measured beginning in the immediate postoperative period on POD0 (in the PACU) and will continue until the end post operative day 2. Oxygen desaturation is defined when measured SpO2 is less than 88%. Measurements will only be recorded if the desaturation event happens for 20 seconds or longer.
PainOUT score | 24 hours post operative discharge, 48 hours post operative discharge, 7 days post operative discharge, 90 days post operative discharge, 180 days post operative discharge
  The severity of post-surgical pain by collecting data on pain intensity, interference with daily activities, and other related factors. Questionnaire uses multiple scales from 0 (none/not at all) to 10 (extreme/severe), percentages 0-100% for amount of pain relief, and "yes" or "no" questions. Higher scores will mean worse outcomes except for pain relief questions which are focused around how much pain relief they felt.
DN4 score | 24 hours post operative discharge, 48 hours post operative discharge, 3 months post operative discharge, 6 months post operative discharge
  DN4 questionnaire to assess neuropathic pain on POD1, 2, 90 and 180. The DN4 questionnaire is a series of Yes or No questions that revolves around the characteristics that may suggest the presence or development of neuropathic conditions/pain.
Opioid-Related Symptom Distress (ORSDS) Scale | 24 hours post operative discharge, 48 hours post operative discharge
  ORSDS questionnaire to assess opioid-related side effects on POD1 and 2. The questionnaire has multiple Yes or No questions, as well as a wording scale from "no side effect" to "almost consistently". Better outcomes will be constant with "no side effect" reported.
Non-opioid analgesic consumption | 24 hours post operative discharge, 48 hours post operative discharge, 7 days post operative discharge
  Patient consumption of non-opioid analgesics from PACU entry through POD7
Sleep disturbance | Post operative day 0 (beginning in the PACU)- 48 hours post operative discharge
  Sleep disturbance via acitgraphy measurement using the ActiGraph wGT3X-BT activity monitor

CONTACTS AND LOCATIONS:
Overall Officials: Kethy Jules-Elysee, M.D., Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article after de-identification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an Independent review committee ("learned intermediary") identified for this purpose and who have signed a DUA.